CLINICAL TRIAL: NCT02582099
Title: Comparison of the Efficacy and Complication of Gentamicin and Normal Saline Nasal Irrigation in Chronic Rhinosinusitis and Recurrent Sinusitis : a Double Blind Randomized Control Trial
Brief Title: The Efficacy and Complication of Gentamicin Nasal Irrigation in Chronic Rhinosinusitis and Recurrent Sinusitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Department of Pediatrics Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 271/2555(EC1)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gentamicin (Active Comparator): Gentamicin nasal irrigation in chronic rhinosinusitis amount 20 ml each pernostril
  Interventions: Drug: Gentamicin nasal irrigation
- Normal saline (Placebo Comparator): Normal saline nasal irrigation in chronic rhinosinusitis amount 20 ml each pernostril
  Interventions: Drug: Normal saline nasal irrigation

INTERVENTIONS:
Drug: Gentamicin nasal irrigation — Nasal wash with gentamicin solution
  Arms: Gentamicin
Drug: Normal saline nasal irrigation — Nasal wash with normal saline solution
  Arms: Normal saline

SUMMARY:
Topical antibiotic therapy in patients with refractory sinusitis has been shown to improve symptoms, quality of life, and mucosal aspect. In pediatrics allergy clinic at Siriraj hospital since 2006 use Gentamicin nasal irrigation for chronic rhinosinusitis.There have been no prospective studies in gentamicin irrigation in chronic rhinosinusitis.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is characterized by symptoms > 12 weeks.Two or more symptoms one of which should be either nasal blockage /obstruction/congestion or nasal discharge (anterior/posterior nasal drip): facial pain/pressure reduction or loss of smell).

Mainstay of treatment are medical and surgical treatment ( ATB, adenoidectomy, ESS) Adjunctive treatment : normal saline nasal irrigation, nasal corticosteroids, nasal decongestants, mucolytics. Nasal lavage with Mupirocin represent an effective and well tolerated alternative treatment of surgically recalcitrant chronic rhinosinusitis. Gentamicin irrigation should be helpful in chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic rhinosinusitis and/or recurrent acute/subacute sinusitis patients who were followed in pediatrics allergy clinic at Siriraj hospital between December 4, 2012, and December 3, 2016

Exclusion Criteria:

1. Patients who used antibiotic prophylaxis within within 1 year before and 6 months after started gentamicin nasal irrigation
2. Patients received IVIG within 1 year before and 6 months after started gentamicin nasal irrigation
3. Patients received IT within 1 year before and 6 months after started gentamicin nasal irrigation
4. Patients underwent endoscopic sinus surgery within 1 year before and 6 months after started gentamicin nasal irrigation
5. Patient who have mental retardation
6. Patient who have aminoglycosides hypersensitivity reactions
7. Pregnancy women and Lactation period
8. Patient who have abnormal hearing test before started gentamicin nasal irrigation
9. Patient who have chronic rhinosinusitis with nasal polyp

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of sinusitis | During 1 year after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand